CLINICAL TRIAL: NCT06689579
Title: Prospective Randomised Controlled Trial of Unipolar vs Bipolar Hemiarthroplasty for Patients With an Intracapsular Hip Fracture
Brief Title: Unipolar vs Bipolar Hemiarthroplasty for Hip Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC: 13/SS/0186 IRAS139897
Record Dates: First submitted 2016-03-21; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unipolar (Experimental): Unipolar hemiarthroplasty used for treatment of intracapsular hip fracture
  Interventions: Device: Unipolar hemiarthroplasty
- Bipolar (Active Comparator): Bipolar hemiarthroplasty used for treatment of intracapsular hip fracture
  Interventions: Device: Bipolar hemiarthroplasty

INTERVENTIONS:
Device: Unipolar hemiarthroplasty
  Other Names: C Stem AMT Unipolar Hemi Arthroplasty DePuy Synthes
  Arms: Unipolar
Device: Bipolar hemiarthroplasty
  Other Names: C Stem AMT Bipolar Hemi Arthroplasty DePuy Synthes
  Arms: Bipolar

SUMMARY:
The purpose of this study is to determine whether significant functional benefits are seen in patients who have a bipolar hemiarthroplasty as treatment for hip fracture compared to those who have a unipolar hemiarthroplasty.

DETAILED DESCRIPTION:
Proposed study design

Randomized controlled trial of unipolar vs bipolar hip hemiarthroplasty for intracapsular fracture of the femoral neck

The trial will be conducted in accordance with the GCP (Good Clinical Practice) guidelines and will be reported in line with the CONSORT statement

Study Centre

The Royal Infirmary of Edinburgh admits 1000 patients a year with a hip fracture; the largest number in any one centre in Scotland. Of these, 500 have intracapsular fractures, which is the type addressed in this study. Some patients will be better suited to a total hip replacement (5-10% of this group), and others may refuse to consent to the trial (previous experience has suggested a rate of 15-20%). Investigators therefore expect just over 300 patients to be recruitable each year, and so plan to allow up to two years for recruitment, and two years to complete follow up of the last patient

Brief Study Method

1. Patients will be identified as requiring a hemiarthroplasty for an intracapsular fracture of the femoral neck
2. Patients will be asked to consent to recruitment to study. Consent by attorney or nearest relative for patients with cognitive impairment
3. Surgery performed via anterolateral approach on standard trauma list. Standard cemented stem implanted.
4. Patient randomized in theatre to receive a unipolar or bipolar hemiarthroplasty head.
5. Tantalum beads will be implanted within the bone of the femur and pelvis (not the hip joint) by a consultant surgeon investigator when operating or assisting personally. These will not implanted where an unsupervised trainee is performing surgery. Fifty patients in each group will have these implants.
6. Patients undergo standard rehabilitation: physiotherapy, occupational therapy and geriatrician services as required.
7. Standard pre-op, post-op and one-year and two-year plain pelvic radiographs will be obtained.
8. Subset of patients: Fifty patients who have received a bipolar hemiarthroplasty will be asked to undergo one additional x-ray of the hip at two years to assess the function of the device.
9. Functional assessment: patients will undergo the Timed up-and-go (TUG) test, physiological measurements of hip muscle recruitment and function, and standardized questionnaires (SF12 and Harris Hip score).

Power analysis and number of patients

200 patients in each arm of study (total 400) allowing for expected 27% mortality at one year.

DMC (Data Monitoring Committee)

A data monitoring committee will review the results during the study period to allow the project to be terminated if statistical significance is reached or if there are any untoward events.

ELIGIBILITY:
Inclusion Criteria

* Patients admitted with an intracapsular fracture of the femoral neck who are suitable for a hemiarthroplasty.

Exclusion Criteria

* Patients deemed suitable for a total hip arthroplasty, patients with a high energy fracture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-10-14 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Pain | 1 year
  visual analogue scale pain score ( on a 10cm baseline fro 'no pain' to 'worst pain imaginable'

SECONDARY OUTCOMES:
Pain | 2 years
  visual analogue scale pain score ( on a 10cm baseline fro 'no pain' to 'worst pain imaginable'
Function | 1 year
  as assessed by 'timed up and go test',
Radiographic assessment | 1 year
  year evidence of acetabular erosion measured with radiostereometric assessment (RSA)
Complications | intraoperative
  duration of surgery (minutes)
Function | 1 year
  physical examination of range of motion
Function | 2 years
  physical examination of range of motion
Function and self care | 1 year
  Barthel Index
Function and self care | 2 years
  Barthel Index
Function and general health | 1 year
  Short form 12
Function and general health | 2 years
  Short form 12
Function | 1 year
  Harris Hip Score
Function | 2 years
  Harris Hip Score
Complications | up to 2 years
  presence of surgical site infection
complications | up to 2 years
  Deep venous thorombosis
complication | up to 2 years
  Periprosthetic fracture
Complication | up to 2 years
  prosthesis dislocation
Complication | up to 2 years
  implant failure
complication | up to 2 years
  repoeration any cause
Complication | up to 2 years
  death
Function | 2 years
  as assessed by 'timed up and go test',

CONTACTS AND LOCATIONS:
Overall Officials: Leela Biant, MD, MBBS, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, Lothian, United Kingdom